CLINICAL TRIAL: NCT07120399
Title: Investigation of the Incidence of Postoperative Chronic Pain in Children Aged 8 to 17 Years
Brief Title: Postoperative Chronic Pain in Children Aged 8 to 17
Status: Not yet recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Onur ERDEM, Research Assistant Doctor, Kocaeli University
Other Study IDs: GOKAEK-2025/06/39
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Chronic Pain
Keywords: Pain; Postoperative Chronic Pain; Quality of Life
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative pediatric patients aged 8-17: Children aged 8 to 17 years who have undergone surgery and voluntarily agree to participate in the study for a period of six months will be included.
  To evaluate pain intensity, the Numeric Rating Scale (NRS) will be utilized, while the Pediatric Quality of Life Inventory 4.0 (PedsQL) will be used to assess quality of life.
  The assessment parameters will be administered at multiple time points: in the preoperative period, at discharge, and on postoperative day 7, as well as at 1 month, 3 months, and 6 months following surgery.

SUMMARY:
The objective of this study is to assess the incidence of chronic postoperative pain in pediatric patients aged 8 to 17 years following surgical procedures. Furthermore, it seeks to identify potential risk factors contributing to the development of such pain and to evaluate its long-term implications.

DETAILED DESCRIPTION:
Children aged 8 to 17 years who have undergone surgery at Kocaeli University Faculty of Medicine and voluntarily agree to participate in the study for a duration of six months will be included.

Children with speech or communication disorders, those who experience postoperative complications, those with psychiatric or neurological conditions, or those with a history of chronic or long-term pain will be excluded from the study.

The participants and their families will be informed about the purpose of the study, the procedures to be followed, the duration of the study, and any potential risks. Written informed consent will be obtained from the parents of all participants. In addition, participants will be asked to complete the informed consent form.

Each participant will be asked to allocate approximately 15 minutes to complete the questionnaires and assessment tools used in the study.

Data such as age, gender, weight, height, ASA score, medical and surgical history, type of surgery, incision size, surgical site, duration of surgery, type of anesthesia and analgesia used, medication doses, intraoperative anesthesia records, length of hospital stay, and any surgical complications will be recorded.

To assess pain intensity, the Numeric Rating Scale (NRS) will be used, and to evaluate quality of life, the Pediatric Quality of Life Inventory 4.0 (PedsQL), which has a validated Turkish version, will be utilized.

These assessment tools will be administered at the following time points: preoperative period, at discharge, and on postoperative day 7, as well as at 1 month, 3 months, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Undergoing a surgical procedure under anesthesia at our hospital
* Availability of complete patient data for a 6-month postoperative follow-up period

Exclusion Criteria:

* Presence of speech or communication disorders
* Development of postoperative complications
* Undergoing any additional surgical procedure for any reason during the 6 months follow-up period
* Having diagnosed psychiatric or neurological disorders
* Having a pre-existing history of chronic or long-term pain

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 8 to 17 years who underwent surgical procedures at Kocaeli University
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
The Numeric Rating Scale (NRS) | Six months
  The Numeric Rating Scale (NRS) is a commonly used pain assessment tool that consists of a numerical scale ranging from 0 to 10. On this scale, 0 indicates no pain, 1 to 3 represents mild pain, 4 to 6 indicates moderate pain, 7 to 9 reflects severe pain, and 10 corresponds to unbearable pain. Patients are asked to select the number that best describes the intensity of pain they are experiencing.

SECONDARY OUTCOMES:
The Pediatric Quality of Life Inventory (PedsQL) | Six months
  The Pediatric Quality of Life Inventory (PedsQL) is a tool designed to measure the quality of life in children and adolescents by assessing their physical, emotional, social, and school functioning. It can be used in both healthy individuals and children with chronic health conditions.
  The PedsQL 4.0 consists of a total of 23 items grouped into four subscales: Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items), and School Functioning (5 items). The inventory includes two parallel forms: one for the child and one for the parent.
  The items are rated using a 5-point Likert scale, where:
  0 = Never a problem
  1. = Almost never a problem
  2. = Sometimes a problem
  3. = Often a problem
  4. = Almost always a problem
  Scores are transformed so that higher scores indicate better quality of life. Score ranges are interpreted as follows:
  80-100: Very good quality of life 60-79: Moderate quality of life 40-59: Low quality of life 0-39: Very low quality

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Faculty of Medicine, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No